CLINICAL TRIAL: NCT03162549
Title: CorEvitas Inflammatory Bowel Disease (IBD) Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-IBD-600
Record Dates: First submitted 2017-05-08; First posted 2017-05-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: Pts presenting to enrolling sites across the US are invited to enroll if eligible

SUMMARY:
This prospective, non-interventional research registry is designed to study the comparative effectiveness and comparative safety of approved treatments for IBD in a cohort of patients cared for by gastroenterologists across North America. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
The objective of the CorEvitas Inflammatory Bowel Diseases (IBD) Registry is to create a national cohort of patients with IBD. The diseases under study include Crohn's Disease (CD) and Ulcerative Colitis (UC). Data collected will be used to better characterize the natural history of the disease and to extensively evaluate the effectiveness and safety of medications approved for the treatment of IBD. This will be done through the standardized collection of validated patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the prevalence and incidence of comorbidities and adverse events, medication utilization patterns, and patient productivity measures.

The design is a prospective, non-interventional registry for patients with IBD under the care of a certified gastroenterologist. Longitudinal follow-up data is collected from both patients and their treating gastroenterologist during routine clinical encounters using CorEvitas registry questionnaires. These questionnaires collect data on patient demographics, disease duration, medical history (including all prior and current treatments for IBD), smoking status, alcohol use, disease activity and severity, pain, as well as other clinician- and patient-reported outcomes, comorbidities and adverse events, infections, hospitalizations, and other targeted safety outcomes.

After the enrollment visit, IBD patients and physicians will complete the follow-up questionnaires during regularly scheduled clinical encounters. The goal is to collect data from patients and providers at six month intervals, not to exceed 2 visits in any 12 month period.

Adverse events may be volunteered spontaneously by the subject, or be discovered as a result of general questioning by the Investigator. During all CorEvitas related visits with the Investigator, subjects will be questioned regarding the occurrence of adverse events.

ELIGIBILITY:
ELIGIBILITY CRITERIA∗ To be eligible for enrollment into the CorEvitas IBD Registry, a patient must satisfy all of the inclusion criteria and none of the exclusion criteria listed below.

Inclusion Criteria:

* At least 18 years of age or older.
* Willing and able to provide written consent for participation in the IBD Registry.
* Willing and able to provide Personally Identifiable Information (PII) which includes the following types of personal information at a minimum: full name, date of birth, sex, and home address zip code.
* Diagnosis of one of the following by a gastroenterologist:

  1. Crohn's disease
  2. Ulcerative colitis
* Prevalent users or new /incident users of an approved biologic drug or JAK inhibitor (Tofacitinib) for the treatment of UC or Crohn's disease.

Exclusion Criteria:

• Participating in or planning to participate in a clinical trial (Phase I - III) or a post-marketing study or registry (i.e. phase IV).∆

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the Inflammatory Bowel Disease (IBD) Registry during regularly -scheduled office visits. Selected gastroenterologist are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 2287 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
IBD epidemiology, presentation, natural history, management, and outcomes | Time Frame: A minimum of 10 years from last patient enrolled
  The major clinical outcomes include an assessment of the epidemiology of Inflammatory Bowel Disease; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Disease burden: Harvey-Bradshaw Index | [Time Frame: every 6 months for 10 years]
Disease burden: Fistula History | [Time Frame: every 6 months for 10 years]
Disease burden: Disease Location and Behavior | [Time Frame: every 6 months for 10 years]
Percentage of patients with history of comorbidities | [Time Frame: time frame: at registry enrollment]
Physician reported: Pouchitis | [Time Frame: time frame: every 6 months for 10 years]
Physician reported: Simple Clinical Colitis Activity Index (SCCAI) | [Time Frame: time frame: every 6 months for 10 years]
Physician reported: Mayo Severity Index | [Time Frame: time frame: every 6 months for 10 years]
Physician reported: IBD related extraintestinal manifestations | [Time Frame: time frame: every 6 months for 10 years]
Patient reported: Patient reported: Work productivity and Activity Impairment (WPAI) | [Time Frame: time frame: every 6 months for 10 years]
Patient reported: PROMIS | [Time Frame: time frame: every 6 months for 10 years]

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Greenberg, MD, Study Director — CorEvitas, LLC
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CorEvitas home page — http://www.corevitas.com